CLINICAL TRIAL: NCT03960957
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of a New Dilution and Injection Volume of AbobotulinumtoxinA for the Treatment of Moderate to Severe Glabellar Lines
Brief Title: Efficacy and Safety of a New Dilution and Injection Volume of AbobotulinumtoxinA for the Treatment of Glabellar Lines
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 43USD1805
Record Dates: First submitted 2019-05-21; First posted 2019-05-23 (Actual); Results first posted 2021-05-11 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2021-05

CONDITIONS: Glabellar Frown Lines
MeSH Terms: interventions — abobotulinumtoxinA

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): AbobotulinumtoxinA
  Interventions: Biological: AbobotulinumtoxinA
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: AbobotulinumtoxinA — Treatment of glabellar facial lines with 50 U AbobotulinumtoxinA
  Arms: Experimental
Other: Placebo — Treatment of glabellar facial lines with placebo
  Arms: Placebo

SUMMARY:
An interventional phase 3 study to evaluate efficacy and safety of a new dilution and injection volume of AbobotulinumtoxinA treatment for glabellar lines

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe glabellar lines at maximum frown
* Understands the study requirements and signs an informed consent form

Exclusion Criteria:

* Botulinum toxin treatment in the face within 6 months prior to study treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2019-06-17 (Actual); Primary Completion 2019-09-27 (Actual); Study Completion 2020-04-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Galderma Study Site, Redondo Beach, California
  - Galderma Study Site, San Diego, California
  - Galderma Study Site, Westport, Connecticut
  - Galderma Study Site, Washington D.C., District of Columbia
  - Galderma Study Site, Coral Gables, Florida
  - Galderma Study Site, Atlanta, Georgia
  - Galderma Study Site, St Louis, Missouri
  - Galderma Study Site, Omaha, Nebraska
  - Galderma Study Site, Cincinnati, Ohio
  - Galderma Study Site, Austin, Texas
  - Galderma Study Site, Spring, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experimental | Placebo
Started | 224 | 77
Completed | 216 | 71
Not Completed | 8 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental | Placebo | Total
Number analyzed (Participants) | 224 | 77 | 301
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.7 (11.43) | 42.5 (11.86) | 44.1 (11.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 195 | 69 | 264
  Male | 29 | 8 | 37
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 2 | 11
  White | 205 | 72 | 277
  More than one race | 4 | 0 | 4
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 224 | 77 | 301
Fitzpatrick Skin Type (FST) [Count of Participants; unit: Participants] — Fitzpatrick Skin Type (FST) is a 6 category classification schema for skin color that is a recognized tool for dermatological research that includes human skin pigmentation as a demographic variable.
  FST I: always burns, never tans FST II: usually burns, tans minimally FST III: sometimes mild burn, tans uniformly FST IV: burns minimally, always tans well FST V: very rarely burns, tans very easily FST VI: never burns
  Participants
    FST I | 4 | 1 | 5
    FST II | 59 | 21 | 80
    FST III | 107 | 40 | 147
    FST IV | 45 | 13 | 58
    FST V | 3 | 1 | 4
    FST VI | 6 | 1 | 7

OUTCOME MEASURES:

1. Primary Outcome: Evaluate Composite Responder Rate at Month 1 for a Single Dose of AbobotulinumtoxinA Compared to Placebo
Description: Composite responder is defined as a subject who achieves a score of 0 or 1 and at least 2 grades improvement on both the Investigator Live Assessment (ILA) and the Subject Self Assessment (SSA)
Time Frame: Month 1 after treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental | Placebo
Number analyzed (Participants) | 224 | 77
Participants | 142 | 0

ADVERSE EVENTS:
Time Frame: 24 weeks
Description: While 224 subjects were randomized to study product (i.e. ITT population), 223 subjects were administered the study product (i.e. safety population).
Arm/Group | Experimental | Placebo
All-Cause Mortality (participants affected / at risk) | 0/223 | 0/77
Serious Adverse Events (participants affected / at risk) | 4/223 | 0/77
Other Adverse Events (participants affected / at risk) | 24/223 | 6/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental (N=223) | Placebo (N=77)
Worsening knee pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acute diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Long QT syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Worsening of hemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental (N=223) | Placebo (N=77)
Headache (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 19 (19) | 3 (3)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Eyelid ptosis (Eye disorders) | 3 (3) | 0 (0)
injection site pain (General disorders) | 1 (1) | 2 (2)
Injection site reaction (General disorders) | 1 (1) | 0 (0)
Injection site discomfort (General disorders) | 0 (0) | 1 (1)
sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PIs agree not to present or publish any data or reports collected individually or by subgroup of sites prior to full, initial publication based on all data obtained from all sites.

DOCUMENTS (2):
  • Study Protocol (2019-01-24): https://cdn.clinicaltrials.gov/large-docs/57/NCT03960957/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-29): https://cdn.clinicaltrials.gov/large-docs/57/NCT03960957/SAP_001.pdf